CLINICAL TRIAL: NCT01933100
Title: Comparison of Brown Rice Based-meal or Polished Rice Based-meal or Wheat Based-meal on Functional Constipation in Young Korean Women: A Opened, Clinical Trial
Brief Title: Comparison of Rice Based-meal on Functional Constipation in Young Korean Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CTCF2_2012_RP
Record Dates: First submitted 2013-08-28; First posted 2013-09-02 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Functional Constipation
Keywords: Functional constipation; Brown rice based-meal; Polished rice based-meal; Wheat based-meal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brown Rice Based-Meal (Experimental): Macronutrient composition of experimental diet were carbohydrate 55~70%, protein 7~20%, fat 15~25%, fiber provided by the experimental diet was designed to adequate intake 20g/day for women
  Interventions: Other: Experimental Diet
- Polished Rice Based-Meal (Experimental): Macronutrient composition of experimental diet were carbohydrate 55~70%, protein 7~20%, fat 15~25%, fiber provided by the experimental diet was designed to adequate intake 20g/day for women
  Interventions: Other: Experimental Diet
- Wheat Based-Meal (Experimental): Macronutrient composition of experimental diet were carbohydrate 55~70%, protein 7~20%, fat 15~25%, fiber provided by the experimental diet was designed to adequate intake 20g/day for women
  Interventions: Other: Experimental Diet

INTERVENTIONS:
Other: Experimental Diet — Macronutrient composition of experimental diet were carbohydrate 55~70%, protein 7~20%, fat 15~25%, fiber provided by the experimental diet was designed to adequate intake 20g/day for women

SUMMARY:
This study was conducted to investigate the effects of rice based-meal on functional constipation in young Korean women.

DETAILED DESCRIPTION:
Studies comparing and evaluating the effects of a rice-based diet and a wheat-based diet on bowel movements are insufficient. In summary, efficient measures are needed to help individuals consume enough dietary fiber from natural sources in daily life to improve their bowel movements, rather than to consume a fiber supplements separated or synthesized from a particular natural food. In this study, investigators compare and evaluate the effects and safety of eating rice-based diets (brown rice-based and white rice-based) and a wheat-based diet in terms of bowel health and bowel movements among young women with functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* Age of 19 to 30 years females
* Meet of Rome Ⅲ diagnostic criteria of functional constipation
* Ability to give informed consent

Exclusion Criteria:

* Subject with a history or evidence of clinically significant gastrointestinal, anorectal, hepatic, renal, neurological, pulmonary, endocrine, blood tumor, psychiatric, cardiovascular disease
* Subjects who have a gastrointestinal (GI) disease (Crohn's disease, etc.) that would increase the influence with absorbance medication or a GI surgery excluding appendectomy and hernia surgery
* Known history of moderate to severe hepatic impairment (i.e., serum ALT>1.5×ULN, AST>1.5×ULN)
* Subjects with significant hypersensitivity about brown rice, polished rice, wheat, milk
* Regular ingestion of probiotic products
* Subjects who received certain medications that cause the alteration of bowel movement within the past 2weeks prior to first administration
* Subjects who participated in other clinical investigation within 2 months prior to first administration
* Subject who drink constantly (21 units/week over)
* Subject who are pregnant or breast feeding
* Subject who have irritable bowel syndrome by ROME Ⅲ criteria
* Any significant condition that, in the opinion of the investigator, could interfere with the subject's participation or compliance in the study(i.e., laboratory test and others)

Ages: 19 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Total colon transit time | 0, 28 days from the start of the study
  Hour of total colonic transit

SECONDARY OUTCOMES:
Stool frequency | 0, 28 days from the start of the study
  Frequency of stool(week)
Fecal weight | 0, 28 days from the start of the study
  weight of fecal
Fecal pH | 0, 28 days from the start of the study
  Fecal pH
Fecal lactic acid | 0, 28 days from the start of the study
  Short chain fatty acid(lactic acid)
Fecal butyric acid | 0, 28 days from the start of the study
  Short chain fatty acid
Fecal propionic acid | 0, 28 days from the start of the study
  Short chain fatty acid
Fecal β-glucuronidase | 0, 28 days from the start of the study
  Fecal enzyme
Fecal urease | 0, 28 days from the start of the study
  Fecal enzyme
Fecal β-glucosidase | 0, 28 days from the start of the study
  Fecal enzyme
Bowel movement | 28 days from the start of the study
  The bowel movement questionnire includes the defecation frequency, bowel time, fecal color, degree of difficulty in defecation and abdominal symptom

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No